CLINICAL TRIAL: NCT00811980
Title: The Effects of Linezolid and Vancomycin on Inflammation and Cellular Signaling Vents
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 00392; Pfizer GA5951WK
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Linezolid; Vancomycin

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heathy Subjects
  Interventions: Drug: Linezolid or Vancomycin

INTERVENTIONS:
Drug: Linezolid or Vancomycin — Whole blood samples from healthy subjects will be incubated with MRSA bacterium or bacterial toxins in the presence and absence of either linezolid or vancomycin. Final concentrations will mimic physiologic conditions. Platelets and leukocytes will be isolated and assayed for the presence of absence of activation and pre-mRNA splicing.
  Other Names: Zyvox

SUMMARY:
We will determine if linezolid inhibits cellular activation and production of pro-inflammatory cytokines, providing mechanistic rationale for its clinical efficacy and the justification for further investigations in S. Aureus sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, taking no medications, and not recently hospitalized

Exclusion Criteria:

* Infection (active)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects who consent to donate blood.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
IL-6 | 12 Months
  Measurement of IL-6 release in response to MRSA.

SECONDARY OUTCOMES:
MCP-1 | 12 Months
  Measurement of MCP-1 release in response to MRSA.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Zimmerman, MD, Principal Investigator — University of Utah